CLINICAL TRIAL: NCT07288541
Title: Promoting Positive Emotions in Adolescents Using Positive Event Training: An Indicated Approach (iPET)
Brief Title: Promoting Positive Emotions in Adolescents Using Positive Events Training: An Indicated Approach
Acronym: iPET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Responsible Party: Principal Investigator, Filip Raes, Prof. dr. Filip Raes, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: G051625N
Record Dates: First submitted 2025-11-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Emotional Distress; Anhedonia
Keywords: positive emotions; anhedonia; positive affect regulation; emotional distress; autobiographical thinking
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Events Training (PET) (Experimental)
  Interventions: Behavioral: Positive Events Training (PET)

INTERVENTIONS:
Behavioral: Positive Events Training (PET) — Positive Event Training or PET is a group-based training program combining Memory Specificity Training (MEST; Raes, 2007) and Future Event Specificity Training (FEST; Dutch version of Hallford et al. (2020): Changing the Future: An initial test of Future Specificity Training).

SUMMARY:
Research shows that high positive emotionality is an essential ingredient in building resilience in youngsters, especially those with a vulnerability to develop depressive symptomatology. It may empower them against actual depression and its various long-term adverse outcomes. One way to achieve positive emotions is via the recollection and anticipation of specific positive events. Therefore, to cultivate positive emotions in young people, a user-friendly group training program was developed, translated from basic research findings: Positive Event Training (PET). Through PET, adolescents learn to solidify positive memories and positive plans for the future. In this project, a comprehensive evaluation of PET's efficacy is conducted using a robust methodology with vulnerable youth.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 years (age)
* moderate level of baseline depressive symptoms Exclusion Criteria: /

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Daily-life positive emotions measured via daily diary items at post-training (adapted from Kirtley et al., 2022) | Measured via nine days of daily diaries (2x/day) immediately after the training (i.e., four weeks after the baseline assessment)
  Mean value of four daily diary items (i.e., "How relaxed, content, enthusiast, good do you feel?"), rated on a 0 ("not at all") to 100 ("a lot") rating scale. Higher values represent, higher levels of positive emotions (min = 0, max = 100).
Daily-life positive emotions measured via daily diary items at follow-up (adapted from Kirtley et al., 2022) | Measured via nine days of daily diaries (2x/day) after two/three months of follow-up after the post-training assessment
  Mean value of four daily diary items (i.e., "How relaxed, content, enthusiast, good do you feel?"), rated on a 0 ("not at all") to 100 ("a lot") rating scale. Higher values represent, higher levels of positive emotions (min = 0, max = 100).
Daily-life anhedonia measured via daily diary items at post-training (adapted from Bogaert et al., 2023) | Measured via nine days of daily diaries (2x/day) immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Mean value of three daily diary items tapping into difficulties experiencing consummatory pleasure, anticipatory pleasure and motivational difficulties using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you find it difficult to enjoy yourself?"; "To what extent did you look forward to doing enjoyable things? (reverse-scored), "Conditional: if 0-50 ("not at all - neutral"): Was this because there really weren't any enjoyable things to look forward to, or because they were there but you couldn't really look forward to them?; "How happy did you feel?" (reverse-scored)). Higher score reflects higher levels of anhedonia (min = 0, max = 100).
Daily-life anhedonia measured via daily diary items at follow-up (adapted from Bogaert et al., 2023) | Measured via nine days of daily diaries (2x/day) after two/three months of follow-up after the post-training assessment
  Mean value of three daily diary items tapping into difficulties experiencing consummatory pleasure, anticipatory pleasure and motivational difficulties using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you find it difficult to enjoy yourself?"; "To what extent did you look forward to doing enjoyable things? (reverse-scored), "Conditional: if 0-50 ("not at all - neutral"): Was this because there really weren't any enjoyable things to look forward to, or because they were there but you couldn't really look forward to them?; "How happy did you feel?" (reverse-scored)). Higher score reflects higher levels of anhedonia (min = 0, max = 100).
Daily-life dampening measured via daily diary items at post-training (adapted from Gérardy et al., in preparation; simplified to better fit target group of adolescents) | Measured via nine days of daily diaries (2x/day) immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Mean value of four daily life items to measure mental strategies to reduce the intensity and/or frequency of positive emotions, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you think, "This pleasant feeling won't last"?"; "To what extent did you think, "I don't deserve to feel good"?"; To what extent did you think, "Something might go wrong that will make my good/pleasant feeling go away"?; "To what extent did you think about how difficult it would be if your good/pleasant feeling suddenly disappeared?"). Higher score reflects higher levels of dampening (min = 0, max = 100).
Daily-life dampening measured via daily diary items at follow-up (adapted from Gérardy et al., in preparation; simplified to better fit target group of adolescents) | Measured via nine days of daily diaries (2x/day) after two/three months of follow-up after the post-training assessment
  Mean value of four daily life items to measure mental strategies to reduce the intensity and/or frequency of positive emotions, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you think, "This pleasant feeling won't last"?"; "To what extent did you think, "I don't deserve to feel good"?"; To what extent did you think, "Something might go wrong that will make my good/pleasant feeling go away"?; "To what extent did you think about how difficult it would be if your good/pleasant feeling suddenly disappeared?"). Higher score reflects higher levels of dampening (min = 0, max = 100).
Daily-life savoring measured via daily diary items at post-training (adapted from Gérardy et al., in preparation; simplified to better fit target group of adolescents) | Measured via nine days of daily diaries (2x/day) immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Mean value of two daily life items tapping into the the engagement in attending to, appreciating and enhancing positive experiences, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you allow the good/pleasant feeling to be there and simply let it be?", "To what extent did you try to really focus your attention on the good/pleasant feeling in order to fully experience it and truly enjoy it?"). Higher scores reflect a higher tendency to savor (min = 0, max = 100).
Daily-life savoring measured via daily diary items at follow-up (adapted from Gérardy et al., in preparation; simplified to better fit target group of adolescents) | Measured via nine days of daily diaries (2x/day) after two/three months of follow-up after the post-training assessment
  Mean value of two daily diary items tapping into the the engagement in attending to, appreciating and enhancing positive experiences, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "To what extent did you allow the good/pleasant feeling to be there and simply let it be?", "To what extent did you try to really focus your attention on the good/pleasant feeling in order to fully experience it and truly enjoy it?"). Higher scores reflect a higher tendency to savor (min = 0, max = 100).
Daily-life emotional distress measured via daily diary items at post-training (derived from Bogaert et al., 2023) | Measured via nine days of daily diaries (2x/day) immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Mean value of three daily diary items to measure anxiety, stress and depressed feelings, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "How anxious did you feel?"; "How depressed (down) did you feel?"; "How stressed did you feel?"). A higher score reflects higher levels of emotional distress (min = 0, max = 100).
Daily-life emotional distress measured via daily diary items at follow-up (derived from Bogaert et al., 2023) | Measured via nine days of daily diaries (2x/day) after two/three months of follow-up after the post-training assessment
  Mean value of three daily diary items to measure anxiety, stress and depressed feelings, using a 0-100 Likert scale (0 = "not at all", 100 = "a lot"; items: "How anxious did you feel?"; "How depressed (down) did you feel?"; "How stressed did you feel?"). A higher score reflects higher levels of emotional distress (min = 0, max = 100).

SECONDARY OUTCOMES:
Episodic future thinking features measured via the Episodic Future Thinking Test (EFT-T; Hallford et al., 2019), and single item rating scales per generated event at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  8 cue words in response to which a positive future event is generated, accompanied with single-item rating scales ranging from 1 (not at all) to 9 (very much). In line with the study of Hallford, Yeow, et al. (2020), participants rate the index of detail (IoD), mental imagery (MI), anticipated (AdP) and anticipatory pleasure (AyP), and perceived control (PC) and perceived likelihood of occurrence (PLO) associated with the generated future events on the EFT-T. Higher scores reflect higher levels of the feature of interest (min = 8; max = 72).
Episodic future thinking features measured via the Episodic Future Thinking Test (EFT-T; Hallford et al., 2019), and single item rating scales per generated event at follow-up | Measured after two/three months of follow-up after the post-training assessment
  8 cue words in response to which a positive future event is generated, accompanied with single-item rating scales ranging from 1 (not at all) to 9 (very much). In line with the study of Hallford, Yeow, et al. (2020), participants rate the index of detail (IoD), mental imagery (MI), anticipated (AdP) and anticipatory pleasure (AyP), and perceived control (PC) and perceived likelihood of occurrence (PLO) associated with the generated future events on the EFT-T. Higher scores reflect higher levels of the feature of interest (min = 8; max = 72).
Autobiographical memory features measured via the Autobiographical Memory (AM) Test (AMT; Raes, Williams, & Hermans, 2009) and single item rating scales per generated event at post-training | Measured via self-report scales immediately after the end of the training (i.e., four weeks after the baseline assessment)
  8 cue words in response to which a positive past event is recalled, accompanied with single-item rating scales ranging from 1 (not at all) to 9 (very much). Participants rate the index of detail (IoD), mental imagery (MI), felt and remembered pleasure (FP and RP), associated with the recalled past events on the AMT. Higher scores reflect higher levels of the feature of interest (min = 8; max = 72).
Autobiographical memory features measured via the Autobiographical Memory (AM) Test (AMT; Raes, Williams, & Hermans, 2009) and single item rating scales per generated event at follow-up | Measured after two/three months of follow-up after the post-training assessment
  8 cue words in response to which a positive past event is recalled, accompanied with single-item rating scales ranging from 1 (not at all) to 9 (very much). Participants rate the index of detail (IoD), mental imagery (MI), felt and remembered pleasure (FP and RP), associated with the recalled past events on the AMT. Higher scores reflect higher levels of the feature of interest (min = 8; max = 72).
Positive Affect subscale of the Positive and Negative Affect Schedule Scales (PANAS; Watson et al., 1988) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Positive affect will be assessed via the Positive Affect subscale of the Positive and Negative Affect Schedule Scales (PANAS; Engelen et al., 2006; Watson et al., 1988). The extent to which 10 positive feelings (e.g., "enthusiastic") were experienced is rated on a 5-point scale ranging from 1 (rarely) to 5 (very often), with higher scores reflecting higher positive affect (min = 10, max = 50).
Positive Affect subscale of the Positive and Negative Affect Schedule Scales (PANAS; Watson et al., 1988) at follow-up | Measured via self-report scales after two/three months of follow-up after the post-training assessment
  Positive affect will be assessed via the Positive Affect subscale of the Positive and Negative Affect Schedule Scales (PANAS; Engelen et al., 2006; Watson et al., 1988). The extent to which 10 positive feelings (e.g., "enthusiastic") were experienced is rated on a 5-point scale ranging from 1 (rarely) to 5 (very often), with higher scores reflecting higher positive affect (min = 10, max = 50).
Leuven Anhedonia Scale (LASS, 2nd version; Nelis et al., 2018) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  12 items rated on a 1-5 Likert scale (1 = "This is completely incorrect for me.", 5 = "This is completely correct to me"). A higher total score reflects higher levels of anhedonia (min = 12, max = 60).
Leuven Anhedonia Scale (LASS, 2nd version; Nelis et al., 2018) at follow-up | Measured via self-report scales after two/three months of follow-up after the post-training assessment
  12 items rated on a 1-5 Likert scale (1 = "This is completely incorrect for me.", 5 = "This is completely correct to me"). A higher total score reflects higher levels of anhedonia (min = 12, max = 60).
Dampening measured via the Leuven Exeter Dampening Scale (LEDS, Bogaert et al., 2025) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  The Leuven Exeter Dampening Scale (LEDS, Bogaert et al., 2025) consists of 13 items rated on a 5-point scale ranging from 1 (not at all) to 5 (very often). A higher score reflects a higher dampening tendency (min = 13, max = 65).
Dampening measured via the Leuven Exeter Dampening Scale (LEDS, Bogaert et al., 2025) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  The Leuven Exeter Dampening Scale (LEDS, Bogaert et al., 2025) consists of 13 items rated on a 5-point scale ranging from 1 (not at all) to 5 (very often). A higher score reflects a higher dampening tendency (min = 13, max = 65).
Savoring measured via the Savoring Subscale of the Four-Factor Model of the Abridged Ways Of Savoring Checklist (WOSC) in Response to Everyday Events (Original scale Bryant and Vernoff, 2007; Four-Factor Model Chadwick, 2012) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  The 10 savoring items of the abridged Ways of Savoring Checklist for Adolescents (not yet validated in Dutch) taps into diverse savoring strategies (WOSC; Chadwick, 2012). Items (e.g., "I looked for other people to share it with") are rated on a 7-point scale ranging from 1 (totally disagree) to 7 (totally agree). Higher scores reflect higher levels of engagement in the respective emotion regulation strategy (min = 10, max = 70).
Savoring measured via the Savoring Subscale of the Four-Factor Model of the Abridged Ways Of Savoring Checklist (WOSC) in Response to Everyday Events (Original scale Bryant and Vernoff, 2007; Four-Factor Model Chadwick, 2012) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  The 10 savoring items of the abridged Ways of Savoring Checklist for Adolescents (not yet validated in Dutch) taps into diverse savoring strategies (WOSC; Chadwick, 2012). Items (e.g., "I looked for other people to share it with") are rated on a 7-point scale ranging from 1 (totally disagree) to 7 (totally agree). Higher scores reflect higher levels of engagement in the respective emotion regulation strategy (min = 10, max = 70).
Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  21 items, rated on a 0-3 Likert scale (0 = "Not at all applicable", 3 = "Almost always applicable"). Higher total (subscale) scores reflect higher levels of emotional distress (depressive symptoms, anxious symptoms and stress; min = 0, max = 63).
Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995) at follow-up | Measured via self-report scales after two/three months of follow-up after the post-training assessment
  21 items, rated on a 0-3 Likert scale (0 = "Not at all applicable", 3 = "Almost always applicable"). Higher total (subscale) scores reflect higher levels of emotional distress (depressive symptoms, anxious symptoms and stress; min = 0, max = 63).
Resilience assessed via the short version of the Connor-Davidson Resilience Scale (CD-RISC; Campbell-Sills & Stein, 2007; Connor & Davidson, 2003; translated into Dutch by Danhof-Pont & Schrier, 2006, 2010) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Statements of the Connor-Davidson Resilience Scale (10 items; e.g., "I am able to adapt to change") are rated on a 5-point scale ranging from 1 (not at all) to 5 (very often), with higher scores reflecting higher levels of resilience (min = 10, max = 50).
Daily-life resilience (general) measured via daily diary item at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent did you feel that you were able to handle many things at the same time?", adapted from Martinez-Corts et al., 2015).
Daily-life resilience (in response to stress) measured via daily diary item at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent were you able to cope easily with those feelings of stress?", adapted from Brogly et al., 2024).
Daily-life resilience (in response to stress, using positive emotions) measured via daily diary item at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent did you try to think of something pleasant from the past or the future to cope with that stress?", new item).
Resilience assessed via the short version of the Connor-Davidson Resilience Scale (CD-RISC; Campbell-Sills & Stein, 2007; Connor & Davidson, 2003; translated into Dutch by Danhof-Pont & Schrier, 2006, 2010) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  Statements of the Connor-Davidson Resilience Scale (10 items; e.g., "I am able to adapt to change") are rated on a 5-point scale ranging from 1 (not at all) to 5 (very often), with higher scores reflecting higher levels of resilience (min = 10, max = 50).
Daily-life resilience (general) measured via daily diary item at follow-up | Measured after two/three months of follow-up after the post-training assessment
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent did you feel that you were able to handle many things at the same time?", adapted from Martinez-Corts et al., 2015).
Daily-life resilience (in response to stress) measured via daily diary item at follow-up | Measured after two/three months of follow-up after the post-training assessment
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent were you able to cope easily with those feelings of stress?", adapted from Brogly et al., 2024).
Daily-life resilience (in response to stress, using positive emotions) measured via daily diary item at follow-up | Measured after two/three months of follow-up after the post-training assessment
  Daily diary item rated on a 0-100 Likert (0 = not at all; 100 = a lot), with higher scores reflecting higher daily-life resilience (item: "To what extent did you try to think of something pleasant from the past or the future to cope with that stress?", new item).
Mental wellbeing measured via the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS; Ikink et al., 2012; Stewart-Brown et al., 2009) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  This self-report scale comprises 7 statements (e.g., "I have been feeling relaxed") rated on a 5-point scale ranging from 1 (never) to 5 (always). Higher scores indicate higher self-reported wellbeing (min = 7, max =35).
Mental wellbeing measured via the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS; Ikink et al., 2012; Stewart-Brown et al., 2009) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  This self-report scale comprises 7 statements (e.g., "I have been feeling relaxed") rated on a 5-point scale ranging from 1 (never) to 5 (always). Higher scores indicate higher self-reported wellbeing (min = 7, max =35).
Persistent negative thinking measured via the Persistent and Intrusive Negative Thoughts Scale (PINTS; Magson et al., 2019; 5 items) at post-training | Measured immediately after the end of the training (i.e., four weeks after the baseline assessment)
  This is a 5-item scale measuring the core characteristics of repetitive negative thinking (Magson et al., 2019). The items are answered on a 5-point frequency scale ranging from never (1) to almost always (5). A higher score reflect higher levels of persisitent negative thinking (min = 5, max = 25).
Persistent negative thinking measured via the Persistent and Intrusive Negative Thoughts Scale (PINTS; Magson et al., 2019; 5 items) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  This is a 5-item scale measuring the core characteristics of repetitive negative thinking (Magson et al., 2019). The items are answered on a 5-point frequency scale ranging from never (1) to almost always (5). A higher score reflect higher levels of persisitent negative thinking (min = 5, max = 25).
Common humanity measured via the "Samen mens zijn" scale (Raes & Bogaert, 2025; unpublished) at post-training | Measured immediately after the end of the training (i.e., four weeks after the end of the baseline assessment)
  Self-report scale consisting of 5 items (e.g., "When I go through difficult things, I realize that others also experience tough moments sometimes, just like I do."), rated on a Likertscale from 1 (never or almost never) to 5 (almost always). A higher score reflects higher levels of common humanity (min = 5, max = 25).
Common humanity measured via the "Samen mens zijn" scale (Raes & Bogaert, 2025; unpublished) at follow-up | Measured after two/three months of follow-up after the post-training assessment
  Self-report scale consisting of 5 items (e.g., "When I go through difficult things, I realize that others also experience tough moments sometimes, just like I do."), rated on a Likertscale from 1 (never or almost never) to 5 (almost always). A higher score reflects higher levels of common humanity (min = 5, max = 25).

OTHER OUTCOMES:
Open questions measuring the engagement with the training material, implementation in daily life and general experiences related to the training | Measured after the training (i.e., 4 weeks after the end of the baseline assessment) and at follow-up (i.e., two/three months after the post-training assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Raes, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No
Data can only be accessed by the involved researchers. Anonymized data can be made available at the end of the study, in line with the data management plan and taking into account the faculties' requirements and ethical principles.